CLINICAL TRIAL: NCT03077282
Title: Quality Control and Safety of Prasaprohyai 95%Ethanolic Extract Capsules in Healthy Volunteer
Brief Title: Safety of Prasaprohyai 95%Ethanolic Extract Capsules in Healthy Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thammasat University (Other)
Collaborators: Thai Traditional Medical Knowledge Fund (Other Government)
Responsible Party: Principal Investigator, Miss Nichamon Mukkasombut, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTU-EC-TM-4-137/59
Record Dates: First submitted 2017-02-16; First posted 2017-03-10 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteers
Keywords: Prasaprohyai extract, Healthy volunteers

STUDY DESIGN:
Intervention Model Description: Volunteers will be divided into 2 groups. One will take Prasaprohyai 95% ethanolic extract capsules at a dose of 100 mg three times a day before meals and the other take Prasaprohyai 95% ethanolic extract capsule at a dose of 200 mg 3 times a day before meals for six weeks. After that, they will cease using the drug for 2 weeks (wash out period). All volunteers will be followed up in the third week, sixth week and eighth week to evaluate the safety of the medicines. The researcher will record data such as age, career, BMI, vital signs, signs and symptoms. Safety will be monitored by hematology tests such as liver function test, renal function test, lipid profile and blood sugar.
  The first step in this research will be to study group 1 (100 mg). If it proves safe, the group 2 (200 mg) will be studied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group1 (Experimental): Group1 will take Prasaprohyai 95% ethanolic extract capsules at a dose of 100 mg three times a day before meals (for 6 weeks)
  Interventions: Drug: Prasaprohyai
- group2 (Experimental): Group2 will take Prasaprohyai 95% ethanolic extract capsules at a dose of 200 mg three times a day before meals (for 6 weeks)
  Interventions: Drug: Prasaprohyai

INTERVENTIONS:
Drug: Prasaprohyai — Prasaprohyai 95% ethanolic extract capsules will take three times a day before meals

SUMMARY:
To investigate the safety of Prasaprohyai 95% ethanolic extract at doses of 100 mg and 200 mg for for 6 weeks. (Clinical Trial phase I)

DETAILED DESCRIPTION:
Sample size Group 1 (100mg/meal) = 6 female, 6 male Group 2 (200mg/meal) = 6 female, 6 male

Volunteers will be divided into 2 groups. One will take Prasaprohyai 95% ethanolic extract capsules at a dose of 100 mg three times a day before meals and the other take Prasaprohyai 95% ethanolic extract capsule at a dose of 200 mg 3 times a day before meals for six weeks. After that, they will cease using the drug for 2 weeks (wash out period). All volunteers will be followed up in the third week, sixth week and eighth week to evaluate the safety of the medicines. The researcher will record data such as age, career, BMI, vital signs, signs and symptoms. Safety will be monitored by hematology tests such as liver function test, renal function test, lipid profile and blood sugar.

The first step in this research will be to study group 1 (100 mg). If it proves safe, the group 2 (200 mg) will be studied.

The data gathered will be evaluated using statistical software. The results are in the form of mean ± standard deviation. The study will be planned as repeated measured ANOVA or Friedman's test in order to evaluate differences between groups, accompanied by using paired t-test or Wilcoxon's test in order to evaluate differences within groups. A significance level of p < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age in range 20-60 years old.
* 2) Healthy, or don't have serious medical conditions such as congestive heart disease, liver and renal dysfunction, uncontrolled hypertension, severe asthma, tuberculosis, HIV in the previous month before being recruited in the study, using history taking and complete physical examination and laboratory result.
* 3) Do not taking a medicine constantly.
* 4) Female not pregnant or lactating (non menopause woman will have a pregnancy test. Time since first day of last menstruation 28-35 days).
* 5) Participant and agreement to follow the instructions for 8 weeks.
* 6) Not a participant in another study.

Exclusion Criteria:

* 1) Allergic reactions to Prasaprohyai medications.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Changes of Hematology test | week0, week3, week6 and week8
  All volunteers will receive a hematology test to check renal function, liver function, lipid profile, glucose, complete blood count

SECONDARY OUTCOMES:
Diary note | Everyday until week8 after took Prasaprohyai
  All volunteers will keep a diary of all symptoms and drugs used during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat university, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
safety of Prasaprohyai 95%ethanolic extract capsules in healthy volunteer (liver function test, renal function test, CBC, BP)